CLINICAL TRIAL: NCT02983825
Title: Impact of Continuous Positive Airway Pressure Level on Ventilation/Perfusion Mismatch in Premature Infants: a Phase II Clinical Trial
Brief Title: Impact of CPAP Level on V/Q Mismatch in Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-013910; 825874 (Other: University of Pennsylvania)
Record Dates: First submitted 2016-11-21; First posted 2016-12-06 (Estimated); Results first posted 2020-07-30 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Infant, Premature, Diseases; Respiratory Insufficiency Syndrome of Newborn
Keywords: CPAP; Bronchopulmonary Dysplasia; Ventilator Induced Lung Injury; V/Q mismatch
MeSH Terms: conditions — Infant, Premature, Diseases; Bronchopulmonary Dysplasia; Ventilator-Induced Lung Injury | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Continuous positive airway pressure (CPAP) level changes (Experimental): Protocol guided changes in CPAP level from clinical baseline, with responsiveness in V/Q mismatch guiding subsequent changes; limited to a range of -2 to +3 cm H2O from baseline
  Interventions: Device: Continuous positive airway pressure (CPAP); level changes

INTERVENTIONS:
Device: Continuous positive airway pressure (CPAP); level changes — as per arm description

SUMMARY:
Continuous positive airway pressure (CPAP) is used in premature infants to maintain lungs open and facilitate gas exchange. When ventilation/perfusion (V/Q) mismatch is present, areas of the lung that are open for gas exchange do not match up with the areas of the lung that are receiving blood for gas exchange. This study measure the responsiveness of V/Q mismatch to changes in the amount (or level) of CPAP.

ELIGIBILITY:
Inclusion Criteria:

1. Born at 27-35 weeks gestational age (GA) by best obstetric estimate, determined by the clinical obstetric team during antepartum admission.
2. Age limits: 24 hours of age - 35 weeks corrected gestational age.
3. On continuous CPAP support between 4-8 cm H2O for greater than 24 hours, as document on the bedside infant flow sheet.
4. Supplemental oxygen requirement, with a fraction of inspired oxygen (FiO2) 0.25 for at least 2 consecutive hours, as documented on the bedside infant flow sheet.

Exclusion Criteria:

1. Congenital anomalies, as determined by the clinical supervising physician.
2. Current or prior air leak syndrome, as determined by the clinical supervising physician.

Ages: 24 Hours to 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-07-08 (Actual); Study Completion 2020-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Bamat, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (3):
- United States (3):
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Pennsylvania Hosptital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bamat NA, Orians CM, Abbasi S, Morley CJ, Ross Russell R, Panitch HB, Handley SC, Foglia EE, Posencheg MA, Kirpalani H. Use of ventilation/perfusion mismatch to guide individualised CPAP level selection in preterm infants: a feasibility trial. Arch Dis Child Fetal Neonatal Ed. 2023 Mar;108(2):188-193. doi: 10.1136/archdischild-2022-324474. Epub 2022 Sep 14. PMID 36104165

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Continuous Positive Airway Pressure (CPAP) Level Changes
Started | 12 (Of 21 enrolled subjects, 9 became ineligible for between consent and intervention)
Completed | 9 (Of 12 subjects starting intervention, 3 met specified stopping critieria)
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Continuous Positive Airway Pressure (CPAP) Level Changes
Number analyzed (Participants) | 12
Age, Continuous [Median (Inter-Quartile Range); unit: days] | 19 [16 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 12
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Ventilation/Perfusion Mismatch
Description: Measured by non-invasive computerized technique based on curvilinear characteristics generated by a best-fit curve connecting the fractional inspired oxygen and corresponding peripheral oxygen saturation pairs; measured as difference in degree of right-shift between baseline and "best" CPAP
Time Frame: variable; up to 2 hours
Measure: Median (Inter-Quartile Range); unit: difference in right shift (kPa)
Arm/Group | Continuous Positive Airway Pressure (CPAP) Level Changes
Number analyzed (Participants) | 9
difference in right shift (kPa) | 1.2 [0 to 3.2]
Statistical Analysis 1: Comparison: Continuous Positive Airway Pressure (CPAP) Level Changes; Within subject repeat analysis; V/Q mismatch (measured as degree of right shift in kPa) baseline vs "best" CPAP; Test type: Superiority — Wilcoxon signed-rank test for nonparametric matched-pairs; p = 0.02, Sign test

2. Secondary Outcome: Best CPAP Level
Description: Defined as the lowest CPAP level associated with an improvement greater than 5% in V/Q mismatch relative to the preceding CPAP level
Time Frame: variable, up to 2 hours
Measure: Median (Inter-Quartile Range); unit: cm H2O
Arm/Group | Continuous Positive Airway Pressure (CPAP) Level Changes
Number analyzed (Participants) | 9
cm H2O | 7 [7 to 8]

ADVERSE EVENTS:
Time Frame: 48 hours after intervention
Description: Adverse event monitoring limited to air leak syndromes (pneumothorax, pulmonary interstitial emphysema, pneumomediastinum; as determined by the clinical supervising physician during routine clinical care) and respiratory deterioration, defined as an increase in baseline FiO2 greater than 0.10 in the 48 hour following the study intervention,
Arm/Group | Continuous Positive Airway Pressure (CPAP) Level Changes
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-20): https://cdn.clinicaltrials.gov/large-docs/25/NCT02983825/Prot_SAP_001.pdf